CLINICAL TRIAL: NCT02419274
Title: The All Age Asthma Cohort (ALLIANCE) of the German Center for Lung Research (DZL), Adult Arm
Brief Title: Adult Arm of DZL All Age Asthma Cohort (ALLIANCE)
Acronym: ALLIANCE
Status: Recruiting | Type: Observational
Sponsor: LungenClinic Grosshansdorf (Other)
Collaborators: German Center for Lung Research (Other); Research Center Borstel (Other)
Responsible Party: Sponsor
Other Study IDs: DZL-GHD-ERA
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: asthma; phenotype; childhood; adulthood
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples With DNA — Collection of blood, nasal secretions, sputum and exhaled breath, such as pharyngeal and nasopharyngeal swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
Deep Phenotyping of adult asthma patients:

* severity from mild to severe
* both atopic and non-atopic
* both childhood and adult onset
* both smokers and non-smokers
* corresponding pediatric cohort (Pediatric Arm of DZL All Age Asthma Cohort) with equivalent SOPs regarding collection of biomaterial and clinical data incl. lung function, further processing of biomaterial and further analyses

DETAILED DESCRIPTION:
The clinical heterogeneity of asthma patients has been increasingly recognised within the last years. Recent studies and articles highlighted the idea of asthma not beeing a single disease but rather a unifying term for multiple phenotypes. Phenotype in this sense is defined as the combination of observable properties of an organism, that are produced by the interactions of a genotype and the environment. In contrast, endotype describes a specific underlying pathophysiological pathway. Linking asthma phenotypes and endotypes in a system biological approach is an important research goal in order to develop targeted therapy, especially for severe asthma.

The advantage the investigators' cohort provides is the collaboration with an equivalent pediatric cohort. In this setting questions regarding disease onset, exacerbation and chronicity can be posed and worked with in a comprehensive manner.

ELIGIBILITY:
Inclusion Criteria:

* Proven Diagnosis according to current GINA Guideline (2014)
* Ability to read and understand German
* Ability to understand and agree to informed consent

Exclusion Criteria:

* History of respiratory tract infection within the last 4 weeks before inclusion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthma of all severity grades, both allergic and non-allergic. Age of Onset childhood and adulthood. Smokers and non-smokers.
  Proven Asthma according to current GINA Guidelines (2014)
  Healthy Control Group.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-03; Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Defining clinical asthma phenotypes by combining clinical, lung function and biomaterial data | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaus F Rabe, MD PhD, Principal Investigator — LungenClinic Grosshansdorf, Grosshansdorf, Germany; Susanne Krauss-Etschmann, PhD, Principal Investigator — Research Center Borstel, Borstel, Germany
Locations (1):
- LungenClinic Grosshansdorf, Großhansdorf, Germany

REFERENCES:
- [Background] Wenzel SE. Asthma phenotypes: the evolution from clinical to molecular approaches. Nat Med. 2012 May 4;18(5):716-25. doi: 10.1038/nm.2678. PMID 22561835
- [Background] Anderson GP. Endotyping asthma: new insights into key pathogenic mechanisms in a complex, heterogeneous disease. Lancet. 2008 Sep 20;372(9643):1107-19. doi: 10.1016/S0140-6736(08)61452-X. PMID 18805339
- [Derived] Habener A, Grychtol R, Gaedcke S, DeLuca D, Dittrich AM, Happle C, Abdo M, Watz H, Pedersen F, Konig IR, Thiele D, Kopp MV, von Mutius E, Bahmer T, Rabe KF, Meyer-Bahlburg A, Hansen G; ALLIANCE Study Group as part of the German Center for Lung Research (DZL); Fuchs O, Roesler B, Welchering N, Kohistani-Greif N, Kurz J, Landgraf-Rauf K, Laubhahn K, Maison N, Liebl C, Schaub B, Ege M, Illi S, Hose A, Zeitlmann E, Berbig M, Marzi C, Schauberger C, Zissler U, Schmidt-Weber C, Ricklefs I, Diekmann G, Liboschik L, Voigt G, Sultansei L, Weckmann M, Nissen G, Kirsten AM, Waschki B, Herzmann C, Biller H, Gaede KI, Bovermann X, Steinmetz A, Husstedt BL, Nitsche C, Veith V, Szewczyk M, Brinkmann F, Malik A, Schwerk N, Dopfer C, Price M, Jirmo AC, Liu B, Calveron MR, Weber S, Foth S, Skevaki C, Renz H, Meyer M, Schildberg T, Rietschel E, van Koningsbruggen-Rietschel S, Alcazar M. IgA+ memory B-cells are significantly increased in patients with asthma and small airway dysfunction. Eur Respir J. 2022 Nov 3;60(5):2102130. doi: 10.1183/13993003.02130-2021. Print 2022 Nov. PMID 35595320
- [Derived] Ronnow SR, Sand JMB, Staunstrup LM, Bahmer T, Wegmann M, Lunding L, Burgess J, Rabe K, Sorensen GL, Fuchs O, Mutius EV, Hansen G, Kopp MV, Karsdal M, Leeming DJ, Weckmann M; ALLIANCE Study Group as part of the German Center of Lung Research (DZL). A serological biomarker of type I collagen degradation is related to a more severe, high neutrophilic, obese asthma subtype. Asthma Res Pract. 2022 Apr 13;8(1):2. doi: 10.1186/s40733-022-00084-6. PMID 35418159
- [Derived] Maison N, Omony J, Illi S, Thiele D, Skevaki C, Dittrich AM, Bahmer T, Rabe KF, Weckmann M, Happle C, Schaub B, Meyer M, Foth S, Rietschel E, Renz H, Hansen G, Kopp MV, von Mutius E, Grychtol R; ALLIANCE Study Group; ALLIANCE Study Group; Fuchs O, Roesler B, Welchering N, Kohistani-Greif N, Kurz J, Landgraf-Rauf K, Laubhahn K, Liebl C, Ege M, Hose A, Zeitlmann E, Berbig M, Marzi C, Schauberger C, Zissler U, Schmidt-Weber C, Ricklefs I, Diekmann G, Liboschik L, Voigt G, Sultansei L, Nissen G, Konig IR, Kirsten AM, Pedersen F, Watz H, Waschki B, Herzmann C, Abdo M, Biller H, Gaede KI, Bovermann X, Steinmetz A, Husstedt BL, Nitsche C, Veith V, Szewczyk M, Brinkmann F, Malik A, Schwerk N, Dopfer C, Price M, Jirmo AC, Habener A, DeLuca DS, Gaedcke S, Liu B, Calveron MR, Weber S, Schildberg T, van Koningsbruggen-Rietschel S, Alcazar M. T2-high asthma phenotypes across lifespan. Eur Respir J. 2022 Sep 29;60(3):2102288. doi: 10.1183/13993003.02288-2021. Print 2022 Sep. PMID 35210326
- [Derived] Weckmann M, Bahmer T, Sand JM, Rank Ronnow S, Pech M, Vermeulen C, Faiz A, Leeming DJ, Karsdal MA, Lunding L, Oliver BGG, Wegmann M, Ulrich-Merzenich G, Juergens UR, Duhn J, Laumonnier Y, Danov O, Sewald K, Zissler U, Jonker M, Konig I, Hansen G, von Mutius E, Fuchs O, Dittrich AM, Schaub B, Happle C, Rabe KF, van de Berge M, Burgess JK, Kopp MV; ALLIANCE Study Group as part of the German Centre for Lung Research (DZL). COL4A3 is degraded in allergic asthma and degradation predicts response to anti-IgE therapy. Eur Respir J. 2021 Dec 9;58(6):2003969. doi: 10.1183/13993003.03969-2020. Print 2021 Dec. PMID 34326188
- [Derived] Holz O, Waschki B, Watz H, Kirsten A, Abdo M, Pedersen F, Weckmann M, Fuchs O, Dittrich AM, Hansen G, Kopp MV, von Mutius E, Rabe KF, Hohlfeld JM, Bahmer T; ALLIANCE Study Group. Breath volatile organic compounds and inflammatory markers in adult asthma patients: negative results from the ALLIANCE cohort. Eur Respir J. 2021 Feb 11;57(2):2002127. doi: 10.1183/13993003.02127-2020. Print 2021 Feb. PMID 33008938
- [Derived] Fuchs O, Bahmer T, Weckmann M, Dittrich AM, Schaub B, Rosler B, Happle C, Brinkmann F, Ricklefs I, Konig IR, Watz H, Rabe KF, Kopp MV, Hansen G, von Mutius E; ALLIANCE Study Group as part of the German Centre for Lung Research (DZL). The all age asthma cohort (ALLIANCE) - from early beginnings to chronic disease: a longitudinal cohort study. BMC Pulm Med. 2018 Aug 20;18(1):140. doi: 10.1186/s12890-018-0705-6. PMID 30126401
- [Derived] Bahmer T, Waschki B, Schatz F, Herzmann C, Zabel P, Kirsten AM, Rabe KF, Watz H; ERA-Study Group. Physical activity, airway resistance and small airway dysfunction in severe asthma. Eur Respir J. 2017 Jan 4;49(1):1601827. doi: 10.1183/13993003.01827-2016. Print 2017 Jan. No abstract available. PMID 28052957